CLINICAL TRIAL: NCT06176235
Title: The Combination of Teriflunomide and High-dose Dexamethasone vs High-dose Dexamethasone Alone as First-line Treatment for Newly Diagnosed Adult Primary Immune Thrombocytopenia (ITP): A Prospective, Multicenter, Randomized Trial
Brief Title: Teriflunomide Plus High-dose Dexamethasone as First-line Treatment in Newly Diagnosed Primary Immune Thrombocytopenia
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Trial withdrawn due to substantial protocol amendments invalidating the original design. With no participants enrolled, this aligns with WHO-ICTRP guidelines. Recruitment has ceased, and the revised protocol has been re-registered as NCT07065968.
Sponsor: Peking University People's Hospital (Other)
Collaborators: Beijing Luhe Hospital (Other); Chinese PLA General Hospital (Other); Navy General Hospital, Beijing (Other); Beijing Hospital (Other Government); Beijing Friendship Hospital (Other); Peking University First Hospital (Other); Peking University Third Hospital (Other); China-Japan Friendship Hospital (Other); Beijing Tsinghua Changgeng Hospital (Other)
Responsible Party: Principal Investigator, Xiao Hui Zhang, Vice president of Peking Univeristy Institute of Hematology, Peking University People's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PKU-TFITP-03
Record Dates: First submitted 2023-12-09; First posted 2023-12-19 (Actual); Last update posted 2025-08-11 (Actual); Status verified 2025-08

CONDITIONS: Immune Thrombocytopenia
Keywords: Teriflunomide; Dexamethasone
MeSH Terms: conditions — Purpura, Thrombocytopenic, Idiopathic | interventions — teriflunomide; Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Teriflunomide plus Dexamethasone (Experimental): Oral Teriflunomide was given at a dose of 7 mg once daily for 24 weeks and dexamethasone was given at a dose of 40mg, orally, once per day for 4 consecutive days (Days 1, 2, 3, and 4). Nonresponsive participants with platelets less than 20 x10^9/L or with active bleeding were allowed to repeat the 4-day course of dexamethasone treatment.
  Interventions: Drug: Teriflunomide; Drug: Dexamethasone
- Dexamethasone (Active Comparator): Dexamethasone was given at a dose of 40mg, orally, once per day for 4 consecutive days (Days 1, 2, 3, and 4). Participants in this treatment arm who failed to achieve a sustained response and had a platelet count of less than 20 x 10^9/L or with active bleeding were also allowed to repeat the 4-day course of dexamethasone treatment.
  Interventions: Drug: Dexamethasone

INTERVENTIONS:
Drug: Teriflunomide — Teriflunomide 7 mg orally once daily for 24 weeks. Dose adjustments were made throughout the study based on individual platelet counts.
  Other Names: AUBAGIO
  Arms: Teriflunomide plus Dexamethasone
Drug: Dexamethasone — Dexamethasone 40 mg orally once daily for four consecutive days (the 4-day course of dexamethasone was repeated in the case of lack of response by day 14).

SUMMARY:
A randomized, open-label, multicenter study to compare the efficacy and safety of teriflunomide plus high-dose dexamethasone compared to high-dose dexamethasone monotherapy for the first-line treatment of adults with newly diagnosed primary immune thrombocytopenia (ITP).

DETAILED DESCRIPTION:
This is a parallel-group, multicenter, randomized controlled trial of 132 adults with ITP in China. Patients were randomized to teriflunomide plus high-dose dexamethasone and high-dose dexamethasone monotherapy group. Patients who do not respond to dexamethasone may receive another cycle of high-dose dexamethasone therapy within 2 weeks. Platelet count, bleeding, and other symptoms were evaluated before and after treatment. Adverse events are also recorded throughout the study.

ELIGIBILITY:
Inclusion Criteria:

1. Newly diagnosed, treatment naïve ITP patients
2. Patients with a platelet count <30,000/μL or a platelet count <50,000/μL with bleeding manifestations at the enrollment;
3. Willing and able to sign written informed consent.

Exclusion Criteria:

1. Received first-line and second-line ITP-modifying therapy (any previous dose of corticosteroids or other immune-suppressive agents);
2. Received chemotherapy or anticoagulants or other drugs affecting the platelet counts within 6 months before the screening visit;
3. Active or a history of malignancy;
4. Positive test result for hepatitis B virus (HBV), hepatitis C virus (HCV), or human immunodeficiency virus (HIV);
5. Pregnancy or lactation;
6. Pre-existing acute or chronic liver disease, or serum alanine aminotransferase (ALT) greater than 2 times the upper limit of normal (ULN);
7. Current or recent (<4 weeks before screening) clinically serious viral, bacterial, fungal, or parasitic infection;
8. A known diagnosis of other autoimmune diseases, established in the medical history and laboratory findings with positive results for the determination of antinuclear antibodies, anti-cardiolipin antibodies, lupus anticoagulant or direct Coombs test;
9. Patients who are deemed unsuitable for the study by the investigator.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-12-19 (Actual); Primary Completion 2024-12-12 (Estimated); Study Completion 2025-05-12 (Estimated)

PRIMARY OUTCOMES:
Sustained response | From the start of study treatment (Day 1) to the end of week 24
  Platelet count over 30,000/μL and at least a 2-fold increase of the baseline count in the absence of bleeding and rescue therapy for at least four of the six visits between weeks 19 and 24.

SECONDARY OUTCOMES:
Overall response | From the start of study treatment (Day 1) to the end of week 24
  Complete response (CR) was defined as platelet count over 100,000/μL and absence of bleeding. Response (R) was defined as platelet count over 30,000/μL and at least a 2-fold increase of the baseline count and absence of bleeding.
Time to response | From the start of study treatment (Day 1) to the end of week 24
  The time from treatment initiation to achieve a CR or a R.
Duration of response | From the start of study treatment (Day 1) to the end of week 24
  The time from the achievement of a complete response or a partial response to the loss of response.
Initial response | From the start of study treatment (Day 1) up to week 4 of treatment
  The number of participants with achievement of CR or R at 4 weeks.
Bleeding events | From the start of study treatment (Day 1) to the end of week 24
  Clinically significant bleeding was assessed using the World Health Organization (WHO) bleeding scale.
Adverse events | From the start of study treatment (Day 1) to the end of follow-up
  Adverse events (AEs) were reported and graded according to the Common Terminology Criteria for Adverse Events (CTCAE), version 5.0.
Health-related quality of life (HRQoL) | From the start of study treatment (Day 1) to the end of week 24
  ITP-patient assessment questionnaire (ITP-PAQ) was used to assess the HRQoL before and after treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Xiao-Hui Zhang, MD, Principal Investigator — Peking University Institute of Hematology, Peking University People's Hospital
Locations (10):
- China (10):
  - Beijing Friendship Hospital, Beijing
  - Beijing Hospital, Beijing
  - Beijing Luhe Hospital, Beijing
  - Beijing Tsinghua Changgeng Hospital, Beijing
  - China-Japan Friendship Hospital, Beijing
  - Chinese PLA General Hospital, Beijing
  - Peking University First Hospital, Beijing
  - Peking University Insititute of Hematology, Peking University People's Hospital, Beijing
  - Peking University Third Hospital, Beijing
  - The Sixth Medical Center of PLA General Hospital, Beijing

IPD SHARING:
Plan to Share IPD: No